CLINICAL TRIAL: NCT04363190
Title: Genomic Instability Associated With Chronic Long Term Exposure to Ionizing Radiation in Vascular Surgeons
Brief Title: Genomic Instability in Vascular Surgeons
Acronym: IRADIENT
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Enrique M. San Norberto, MD, PhD, Chief of Unit, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI-18-967
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Cytogenetic Abnormality; Radiation Exposure
Keywords: Vascular surgery; Endovascular surgery
MeSH Terms: conditions — Chromosome Aberrations | interventions — Cytogenetic Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — peripheral blood sample, to obtain peripheral lymphocytes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases
  Interventions: Diagnostic Test: Cytogenetic analysis
- Controls
  Interventions: Diagnostic Test: Cytogenetic analysis

INTERVENTIONS:
Diagnostic Test: Cytogenetic analysis — 1. FISH study using the UroVysion kit in interphase peripheral lymphocytes, that allows the study of numerical aberrations for chromosomes 3, 7 and 17 and locus 9p21.
  2. G banding study to analyse the whole karyotype study regarding both numerical and structural aberrations during metaphase.
  3. Sister chromatid exchanges (SCE) analysis with bromodeoxyuridine (BrdU) staining for the whole karyotype during metaphase: analizing the proportion of SCE per metaphase (NSM).

SUMMARY:
The past two decades have witnessed the development and growth of the endovascular techniques, however, this new technology is not exempt from risks, since its use requires an ionizing radiation exposure to both patients and surgeons. In this context, the long-term repercussion of this type of chronic exposure to low dose ionizing radiation of the vascular surgeons is still unknown. Although conventional dosimetry is used to monitoring the occupational radiation exposure, it doesn't take into consideration a number of individual variables such as: age, sex, exposure to other carcinogen substances or previous medical history; that may affect the radio-sensibility of each individual. Some studies suggest the use of routine cytogenetic analysis to complement the conventional dosimetry, yet the real genomic effects of chronic low dose ionizing radiation exposure is still unclear and an ideal biodosimetry marker hasn't been described. In this setting, the main objective of the present study was to determine the genomic instability associated to the chronic low dose exposure to ionizing radiation of vascular surgeons versus healthy control patients with no history of radiation exposure.

The secondary endpoints were to determine the impact of demographic and clinical practice activities associated to genomic instability among both groups of patients.

National, observational and transversal case control study of genomic instability among vascular surgeons chronically exposed to low dose ionizing radiation compared to healthy control patients with no previous history of radiation exposure. The peripheral blood samples of the case group were collected from vascular surgeons during the VI International Symposium of Endovascular Surgery. The blood samples were followed by a demographic and endovascular practice questionnaire. On the other hand, the samples for the control group were collected from healthy patients undergoing saphenectomy and/or phlebectomy in our department at Hospital Clínico Universitario de Valladolid. All blood samples were send to the Cancer Investigation Center at Salamanca University where three types of genomic analysis were performed: (1) fluorescence in situ hybridization (FISH) study in interphase for the chromosomes 3, 7 and 17 and locus 9p21; (2) metaphase study with G banding technique; and (3) sister chromatid exchange (SCE) metaphase study.

ELIGIBILITY:
Inclusion Criteria:

Cases

* Vascular surgeons regularly involved in endovascular procedures.
* Over 10 years of endovascular experience.
* Accept to participate in the present study.

Controls:

* Healthy patients undergoing saphenectomy and/or phlebectomy.
* Accept to participate in the present study.

Exclusion Criteria:

Cases:

* Less than 10-year endovascular experience.
* Previous medical history of cancer.
* Have been treated with radiotherapy.
* Have been exposed to ionizing radiation outside the endovascular field.
* Not accept to participate in the present study.

Controls:

* Previous medical history of cancer.
* Have been treated with radiotherapy.
* Have been exposed to ionizing radiation.
* Not accept to participate in the present study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The peripheral blood samples of the case group were collected from vascular surgeons during the VI International Symposium of Endovascular Surgery. The blood samples were followed by a demographic and endovascular practice questionnaire. On the other hand, the samples for the control group were collected from healthy patients undergoing saphenectomy and/or phlebectomy in our department at Hospital Clínico Universitario de Valladolid.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
The differences between cases and controls regarding chromosomal numerical aberrations during interphase using FISH technique | 2 years
  The differences between cases and controls regarding chromosomal numerical aberrations during interphase of chromosomes 3, 7, 17 and locus 9p21.
  The differences between cases and controls regarding chromosomal numerical aberrations during interphase using FISH technique with the UroVysion kit for chromosomes 3, 7, 17 and locus 9p21.
The differences between cases and controls after G banding technique | 2 years
  The differences between cases and controls regarding chromosomal numerical and structural aberrations during metaphase.
The differences between cases and controls regarding the presence of SCE during metaphase. | 2 years
  The differences between cases and controls regarding the presence of SCE during metaphase.

SECONDARY OUTCOMES:
Demographic variables, in terms of age and sex, regarding the presence of chromosomal aberrations and SCE. | 2 years
  Demographic variables, in terms of age and sex, regarding the presence of chromosomal aberrations and SCE.
The impact of the anatomical region treated as well as the performance of complex aortic endovascular procedures amongst the group of vascular surgeons included in the present study regarding the presence of chromosomal aberrations and SCE. | 2 years
  The impact of the anatomical region treated as well as the performance of complex aortic endovascular procedures amongst the group of vascular surgeons included in the present study regarding the presence of chromosomal aberrations and SCE.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universtario de Valladolid, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mu H, Sun J, Li L, Yin J, Hu N, Zhao W, Ding D, Yi L. Ionizing radiation exposure: hazards, prevention, and biomarker screening. Environ Sci Pollut Res Int. 2018 Jun;25(16):15294-15306. doi: 10.1007/s11356-018-2097-9. Epub 2018 Apr 29. PMID 29705904
- [Result] Jaco JW, Miller DL. Measuring and monitoring radiation dose during fluoroscopically guided procedures. Tech Vasc Interv Radiol. 2010 Sep;13(3):188-93. doi: 10.1053/j.tvir.2010.03.009. PMID 20723835
- [Result] Balter S, Hopewell JW, Miller DL, Wagner LK, Zelefsky MJ. Fluoroscopically guided interventional procedures: a review of radiation effects on patients' skin and hair. Radiology. 2010 Feb;254(2):326-41. doi: 10.1148/radiol.2542082312. PMID 20093507
- [Result] Hertault A, Maurel B, Midulla M, Bordier C, Desponds L, Saeed Kilani M, Sobocinski J, Haulon S. Editor's Choice - Minimizing Radiation Exposure During Endovascular Procedures: Basic Knowledge, Literature Review, and Reporting Standards. Eur J Vasc Endovasc Surg. 2015 Jul;50(1):21-36. doi: 10.1016/j.ejvs.2015.01.014. Epub 2015 Mar 25. PMID 25818982
- [Result] Stecker MS, Balter S, Towbin RB, Miller DL, Vano E, Bartal G, Angle JF, Chao CP, Cohen AM, Dixon RG, Gross K, Hartnell GG, Schueler B, Statler JD, de Baere T, Cardella JF; SIR Safety and Health Committee; CIRSE Standards of Practice Committee. Guidelines for patient radiation dose management. J Vasc Interv Radiol. 2009 Jul;20(7 Suppl):S263-73. doi: 10.1016/j.jvir.2009.04.037. No abstract available. PMID 19560006
- [Result] Wdowiak A, Skrzypek M, Stec M, Panasiuk L. Effect of ionizing radiation on the male reproductive system. Ann Agric Environ Med. 2019 Jun 17;26(2):210-216. doi: 10.26444/aaem/106085. Epub 2019 May 6. PMID 31232047
- [Result] Sunada S, Haskins JS, Kato TA. Sister Chromatid Exchange as a Genotoxic Stress Marker. Methods Mol Biol. 2019;1984:61-68. doi: 10.1007/978-1-4939-9432-8_7. PMID 31267420
- [Result] Wilson DM 3rd, Thompson LH. Molecular mechanisms of sister-chromatid exchange. Mutat Res. 2007 Mar 1;616(1-2):11-23. doi: 10.1016/j.mrfmmm.2006.11.017. Epub 2006 Dec 6. PMID 17157333
- [Result] Miller DL, Vano E, Bartal G, Balter S, Dixon R, Padovani R, Schueler B, Cardella JF, de Baere T; Cardiovscular and Interventional Radiology Society of Europe; Society of Interventional Radiology. Occupational radiation protection in interventional radiology: a joint guideline of the Cardiovascular and Interventional Radiology Society of Europe and the Society of Interventional Radiology. Cardiovasc Intervent Radiol. 2010 Apr;33(2):230-9. doi: 10.1007/s00270-009-9756-7. Epub 2009 Dec 18. No abstract available. PMID 20020300
- [Result] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Result] Boc V, Boc A, Zdesar U, Blinc A. Patients' radiation doses during percutaneous endovascular procedures in arteries of the lower limbs. Vasa. 2019 Mar;48(2):167-174. doi: 10.1024/0301-1526/a000744. Epub 2018 Oct 16. PMID 30322344
- [Result] Dendy PP. Radiation risks in interventional radiology. Br J Radiol. 2008 Jan;81(961):1-7. doi: 10.1259/bjr/15413265. Epub 2007 Nov 26. PMID 18039723
- [Result] Sailer AM, Schurink GW, Bol ME, de Haan MW, van Zwam WH, Wildberger JE, Jeukens CR. Occupational Radiation Exposure During Endovascular Aortic Repair. Cardiovasc Intervent Radiol. 2015 Aug;38(4):827-32. doi: 10.1007/s00270-014-1025-8. Epub 2014 Dec 5. PMID 25476871
- [Result] Patel AP, Gallacher D, Dourado R, Lyons O, Smith A, Zayed H, Waltham M, Sabharwal T, Bell R, Carrell T, Taylor P, Modarai B. Occupational radiation exposure during endovascular aortic procedures. Eur J Vasc Endovasc Surg. 2013 Oct;46(4):424-30. doi: 10.1016/j.ejvs.2013.05.023. Epub 2013 Jul 19. PMID 23871303
- [Result] Kostova-Lefterova DD, Nikolov NN, Stanev SS, Stoyanova BB. Patient doses in endovascular and hybrid revascularization of the lower extremities. Br J Radiol. 2018 Nov;91(1091):20180176. doi: 10.1259/bjr.20180176. Epub 2018 Aug 13. PMID 30028182
- [Result] Ingwersen M, Drabik A, Kulka U, Oestreicher U, Fricke S, Krankenberg H, Schwencke C, Mathey D. Physicians' radiation exposure in the catheterization lab: does the type of procedure matter? JACC Cardiovasc Interv. 2013 Oct;6(10):1095-102. doi: 10.1016/j.jcin.2013.05.012. PMID 24156970
- [Result] Majewska N, Blaszak MA, Juszkat R, Frankiewicz M, Makalowski M, Majewski W. Patients' radiation doses during the implantation of stents in carotid, renal, iliac, femoral and popliteal arteries. Eur J Vasc Endovasc Surg. 2011 Mar;41(3):372-7. doi: 10.1016/j.ejvs.2010.10.018. Epub 2010 Dec 13. PMID 21147004
- [Result] Sigterman TA, Bolt LJ, Snoeijs MG, Krasznai AG, Heijboer R, Schurink GW, Bouwman LH. Radiation Exposure during Percutaneous Transluminal Angioplasty for Symptomatic Peripheral Arterial Disease. Ann Vasc Surg. 2016 May;33:167-72. doi: 10.1016/j.avsg.2015.11.019. Epub 2016 Feb 21. PMID 26902938
- [Result] Stanisic MG, Majewska N, Makalowski M, Juszkat R, Blaszak M, Majewski W. Patient radiation exposure during carotid artery stenting. Vascular. 2015 Apr;23(2):154-60. doi: 10.1177/1708538114540641. Epub 2014 Jun 25. PMID 24966273
- [Result] Neill M, Charles HW, Pflager D, Deipolyi AR. Factors associated with reduced radiation exposure, cost, and technical difficulty of inferior vena cava filter placement and retrieval. Proc (Bayl Univ Med Cent). 2017 Jan;30(1):21-25. doi: 10.1080/08998280.2017.11929515. PMID 28127123
- [Result] Santovito A, Cervella P, Delpero M. Increased frequency of chromosomal aberrations and sister chromatid exchanges in peripheral lymphocytes of radiology technicians chronically exposed to low levels of ionizing radiations. Environ Toxicol Pharmacol. 2014 Jan;37(1):396-403. doi: 10.1016/j.etap.2013.12.009. Epub 2013 Dec 31. PMID 24440812
- [Result] Lee WH, Nguyen PK, Fleischmann D, Wu JC. DNA damage-associated biomarkers in studying individual sensitivity to low-dose radiation from cardiovascular imaging. Eur Heart J. 2016 Oct 21;37(40):3075-3080. doi: 10.1093/eurheartj/ehw206. Epub 2016 Jun 5. No abstract available. PMID 27272147
- [Result] Rosolen DCB, Faria DK, Faria CS, Antonangelo L. Performance of the UroVysion(R) FISH assay for the diagnosis of malignant effusions using two cutoff strategies. Cancer Med. 2018 May;7(5):1967-1977. doi: 10.1002/cam4.1442. Epub 2018 Mar 25. PMID 29577646